CLINICAL TRIAL: NCT02421107
Title: A Clinical Study to Evaluate the Safety of the GlySure Continuous Intravascular Glucose Monitoring System, and Its Performance in Comparison to Intermittent Blood Glucose Monitoring in Adult Intensive Care Unit Patients
Brief Title: GlySure Acute Care Settings Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: GlySure (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group
Other Study IDs: 2014.02.CE
Record Dates: First submitted 2014-11-03; First posted 2015-04-20 (Estimated); Last update posted 2015-04-20 (Estimated); Status verified 2015-04

CONDITIONS: Adult Intensive Care Patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- all patients (Other): all patients
  Interventions: Other: Glysure CGM; Other: iStat intermittent testing

INTERVENTIONS:
Other: Glysure CGM
Other: iStat intermittent testing

SUMMARY:
The company who have developed the GlySure product have previously carried out a study to be able to show that the GlySure system is accurate in measuring blood sugar (glucose) levels. This was done with patients in the intensive care unit (ICU) after heart surgery.

The company now want to confirm that the GlySure product is accurate at measuring blood glucose levels on all patients who stay in the ICU.

This clinical study requires 40 patients and is to check the safety of a continuous Glucose Monitoring System (GlySure) and it's performance in comparison to separate individual blood glucose testing using a hand held blood tester called i-STAT. Each patient must be in the study for at least 36 hours.

The main benefit of continuous blood glucose monitoring is that it gives a true picture of the glucose status of a patient and this can potentially help avoid the glucose level dropping too low (hypoglycaemic) or staying too high (hyperglycaemia) as clinicians can intervene based on 'real-time' data on the glucose levels.

In this study patient treatment is not dictated by the data measured during the study. Clinicians are blind to the results on the GlySure monitor.

ELIGIBILITY:
Inclusion Criteria:

1. Patient or legal representative MUST be willing to sign an informed consent document
2. Patient is male or female aged 18 years or above
3. Patient requires a Central Venous Catheter (CVC) to be inserted as part of disease management and treatment
4. Patient is expected to remain in the intensive care unit for at least 36 hours post enrolment to the study

Exclusion Criteria:

1. Patient or legal representative is unable to provide written informed consent
2. Patient who is pregnant
3. Patient who is currently being administered Mannitol and/or may require the administration of Mannitol whilst in the ICU
4. Patient with history of pulmonary embolism (PE)
5. Patient with history of thrombosis
6. Patient with known hyper-coagulation
7. Patient with known history of heparin hypersensitivity
8. Patient with history of heparin induced thrombocytopenia
9. Participation in a clinical study involving an unlicensed pharmaceutical product or device within the 3 months prior to enrolment in this study
10. Patient with known hypersensitivity/allergy to adhesive I.V. dressings such as 3M Tegaderm film or StatLock® devices
11. Patient who is being managed in a cardiac ICU setting after cardiac surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-04; Primary Completion 2015-08 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
safety as assessed by serious adverse events attributed to the study investigational product | 0-7 days
mean absolute relative difference (MARD) % (accuracy) | 0-7 days